CLINICAL TRIAL: NCT03342378
Title: PET-MRI Assessment of Early Tumor Response to Predict Outcomes of HPV-Positive Oropharynx Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: UW17078; 2017-1010 (Other: Institutional Review Board); P50DE026787 (NIH); Protocol Version 1/7/2020 (Other: UW Madison)
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Squamous Cell Carcinoma; Oropharynx Cancer
Keywords: HPV; HPV-positive; Oropharynx Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Oropharyngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oropharynx Cancer Patients: Patients with OPSCC will be treated with comprehensive head and neck RT to 70 Gy in 33 fractions with concurrent weekly cisplatin at 40 mg/m2 and at the University of Wisconsin.
  Interventions: Radiation: Intensity modulated radiotherapy (IMRT); Diagnostic Test: PET-MRI

INTERVENTIONS:
Radiation: Intensity modulated radiotherapy (IMRT) — Intensity modulated radiotherapy (IMRT) will be delivered over 6.5 weeks in 33 daily fractions. Treatments will be initiated on Monday or Tuesday. Missed treatments will be compensated for by delivering an additional BID treatment during the week given at least 6 hours apart OR treating on the Saturday of that week, OR adding to the end of treatment. Gross disease will receive 70 Gy in 2.12 Gy fractions, areas at high-risk for subclinical disease will receive 60 Gy in 1.82 Gy fractions, and areas at low-risk for harboring subclinical disease will receive 56 Gy in 1.70 Gy fractions.
Diagnostic Test: PET-MRI — All imaging data will be acquired using a 3.0T PET-MRI scanner with a standard bore size of 60 cm. Patients will be placed in standard non-ferrous head and neck immobilization devices during PET-MRI to simulate their anticipated positioning during subsequent CT simulation and treatment. A head and neck PET-MRI study will be performed with scan sequences tailored for the site of interest. The PET-MRI exam will take approximately 90 minutes to complete.

SUMMARY:
This proposal explores the novel hypothesis that the variability in outcomes within the Intermediate Risk(IR) HPV-positive Oropharynx Squamous Cell Carcinoma(OPSCC) cohort can be exploited to identify a subpopulation that exhibits outcomes similar to Low Risk (LR) HPV-positive Oropharynx Squamous Cell Carcinoma and therefore would be appropriate candidates for radiation dose de-escalation approaches. Current literature using PET, CT, and MRI as single imaging modalities have identified certain criteria within heterogenous patient populations that are associated with clinical outcomes. Here, the investigators will test the hypothesis that multiparametric analysis of simultaneously-acquired MRI and PET quantitative imaging biomarker data from the primary tumor prior to initiating therapy, after 2 weeks of chemoradiation(CRT), and 3 months following completion of chemoradiation in patients with Intermediate Risk HPV-positive Oropharynx Squamous Cell Carcinoma will generate parametric maps that are predictive of clinical outcome.

Furthermore, the investigators will collect blood samples prior to, during, and after radiation therapy to evaluate whether levels of detected circulating tumor cells correlate with response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-proven diagnosis of squamous cell carcinoma (including papillary squamous cell carcinoma and basaloid squamous cell carcinoma variants) of the oropharynx (tonsil or base of tongue)
* III-IVB (T3N0, T1-3N1, T4aN0-3, T4bN0-3, T1-4N2, T1-4N3) (AJCC 8th edition) based upon the following minimum diagnostic workup:

  * General history and physical examination (including nasolarygopharyngoscopy or indirect mirror exam) by a radiation oncologist or medical oncologist or ENT head and neck surgeon within 8 weeks prior to registration.
  * Diagnostic CT of the neck with IV contrast
  * Chest imaging

    * CXR or CT chest without contrast
* Patient must not have any contraindications to undergoing a 3.0T PET-MRI
* Zubrod Performance Status 0-1 within 2 weeks prior to registration.
* Smoking history defined by pack-years (calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked).
* Negative urine pregnancy test within 2 weeks prior to registration for women of childbearing potential.
* Patient must provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Cancers considered to be from an oral cavity, nasopharynx, hypopharynx, or larynx are excluded. Carcinoma of the neck of unknown primary site origin (even if p16 positive) are excluded.
* Distant metastasis
* Gross total excision of the primary tumor with or without nodal dissection.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years. (For example, carcinoma of the breast, colon or cervix are all permissible if patients are disease free for ≥ 3 years.)
* Prior radiotherapy to the head and neck region that would result in overlap of radiation therapy fields.
* Presence of passive and/or active devices that are not compatible with the 3.0T PET/MR scanner environment. Any person with the following will be excluded: cardiac pacemaker, metal fragments in or around the eye, venous umbrella, permanent eyeliner or permanent artificial eyebrows. Patents with the following potentially non-MRI compatible devices will undergo screening using the standard UWHC MRI screening protocol by trained UWHC personnel: cardiac pacemaker, heart valve replacement, intracranial aneurysm clips, middle ear, eye, joint, or penile implants, joint replacements, implantable hearing aids, neurostimulator devices, insulin pumps, shunts/stents, metal mesh/coil implants; metal plate/pin/screws/wires, or any other metallic implants. Also, patients with anatomical constraints limiting the feasibility of MRI will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with OPSCC will be enrolled on an institutional review board approved clinical trial and treated with comprehensive head and neck RT to 70 Gy in 33 fractions, some with concurrent weekly cisplatin at 40 mg/m2 and at the University of Wisconsin.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Radiographic change in the primary tumor of patients with LR and IR HPV-positive OPSCC using MRI/PET imaging | Pre-treatment (baseline) and following 2-weeks of CRT (approximately 2-3 weeks on study)
  Patients with LR and IR HPV-positive OPSCC will be segregated into favorable and unfavourable cohorts using radiographic change(MRI/PET) in the primary tumor between pre-treatment and intra-treatment. T-stage, N-stage, and pack-years smoking markers will be used as surrogate markers
Radiographic change in the primary largest pathologic lymph node of patients with LR and IR HPV-positive OPSCC using MRI/PET imaging | Pre-treatment (baseline) and following 2-weeks of CRT (approximately 2-3 weeks on study)
  Patients with LR and IR HPV-positive OPSCC will be segregated into favorable and unfavourable cohorts using radiographic change(MRI/PET) in the largest pathologic lymph node between pre-treatment and intra-treatment. T-stage, N-stage, and pack-years smoking markers will be used as surrogate markers

SECONDARY OUTCOMES:
Progression Free Survival | up to 2 years
Absolute volumetric change of the primary tumor | Following 2-weeks of CRT (approximately 2-3 weeks on study)
  The primary tumor response in patients with LR HPV-positive OPSCC and HPV-negative OPSCC will be measured in terms of absolute volumetric change in the tumor following 2 weeks of CRT
Absolute metabolic change of the primary tumor | Following 2-weeks of CRT (approximately 2-3 weeks on study)
  The primary tumor response in patients with LR HPV-positive OPSCC and HPV-negative OPSCC will be measured in terms of absolute metabolic change in the tumor following 2 weeks of CRT
Absolute physiologic change of the primary tumor | Following 2-weeks of CRT (approximately 2-3 weeks on study)
  The primary tumor response in patients with LR HPV-positive OPSCC and HPV-negative OPSCC will be measured in terms of absolute physiologic change in the tumor following 2 weeks of CRT
Absolute volumetric change of involved nodes | Following 2-weeks of CRT (approximately 2-3 weeks on study)
  The nodal response in patients with LR HPV-positive OPSCC and HPV-negative OPSCC will be measured in terms of absolute volumetric change of involved nodes following 2 weeks of CRT
Absolute metabolic change of involved nodes | Following 2-weeks of CRT (approximately 2-3 weeks on study)
  The nodal response in patients with LR HPV-positive OPSCC and HPV-negative OPSCC will be measured in terms of absolute metabolic change of involved nodes following 2 weeks of CRT
Absolute physiologic change of involved nodes | Following 2-weeks of CRT (approximately 2-3 weeks on study)
  The nodal response in patients with LR HPV-positive OPSCC and HPV-negative OPSCC will be measured in terms of absolute physiologic change of involved nodes following 2 weeks of CRT

OTHER OUTCOMES:
Number of Circulating Tumor Cells | Pre-treatment (baseline) and following 2-weeks of CRT (approx. 2-3 weeks on study), 3-months post-treatment (approx. 19-23 weeks on study)
Change in Number of Circulating Tumor Cells Between Time Points | Pre-treatment (baseline) and following 2-weeks of CRT (approx. 2-3 weeks on study), 3-months post-treatment (approx. 19-23 weeks on study)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Kimple, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] Witek ME, Kimple RJ, Avey GD, Burr AR, Chandereng T, Yu M, Hu R, Wieland AM, Labby ZE, Bruce JY, Brower JV, Hartig GK, Harari PM. Prospective Study of PET/MRI Tumor Response During Chemoradiotherapy for Patients With Low-risk and Intermediate-risk p16-positive Oropharynx Cancer. Am J Clin Oncol. 2022 May 1;45(5):202-207. doi: 10.1097/COC.0000000000000910. Epub 2022 Apr 12. PMID 35446279
- See also: UW Carbone Cancer Center Homepage — http://cancer.wisc.edu/